CLINICAL TRIAL: NCT02569775
Title: Outcomes of Autologous Bone Marrow Mononuclear Cells for Cerebral Palsy: A Self-Controlled Clinical Trial
Brief Title: Outcomes of Stem Cells for Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBG 001
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Stem Cells
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cell transplantation (Experimental): 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 3 months afterward
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Bone Marrow Mononuclear Cells — Transplantation of Autologous Bone Marrow Mononuclear Cells

SUMMARY:
The aim of this study is to assess the safety and effectiveness of autologous bone marrow mononuclear stem cells in patients with cerebral palsy.

DETAILED DESCRIPTION:
The aim of this study is to assess the safety and effectiveness of autologous bone marrow mononuclear stem cells in 40 patients with cerebral palsy at Vinmec International Hospital, Hanoi, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy of any types caused by oxygen deprivation.

Exclusion Criteria:

* Epilepsy
* Hydrocephalus with ventricular drain
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Total Score of Gross Motor Function Measure (GMFM)-88 | 3 months and 6 months after transplantation
  GMFM-88
Change in Gross Motor Function Measure (GMFM)-66 Percentile | 3 months and 6 months after transplantation
  GMFM-66 percentile

SECONDARY OUTCOMES:
Change in Muscle tone | 3 months and 6 months after transplantation
  Muscle tone are assessed by Modified Ashworth Scale
Number of adverse events | Through study completion, an average of 6 months
  Examples of adverse events to look for: anaphylaxis, allergy, respiratory distress, fever, infections, vomit, epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD., Study Chair — Vinmec Healthcare System
Locations (1):
- Vinmec International Hospital, Hanoi, Vietnam

REFERENCES:
- [Background] Sharma A, Sane H, Gokulchandran N, Kulkarni P, Gandhi S, Sundaram J, Paranjape A, Shetty A, Bhagwanani K, Biju H, Badhe P. A clinical study of autologous bone marrow mononuclear cells for cerebral palsy patients: a new frontier. Stem Cells Int. 2015;2015:905874. doi: 10.1155/2015/905874. Epub 2015 Feb 18. PMID 25788947
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596
- [Derived] Nguyen LT, Nguyen AT, Vu CD, Ngo DV, Bui AV. Outcomes of autologous bone marrow mononuclear cells for cerebral palsy: an open label uncontrolled clinical trial. BMC Pediatr. 2017 Apr 12;17(1):104. doi: 10.1186/s12887-017-0859-z. PMID 28403842